CLINICAL TRIAL: NCT02122107
Title: Cognition in Older Breast Cancer Survivors: Treatment Exposure, APOE and Smoking History
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: City of Hope Medical Center (Other); The New School for Social Research (Other)
Responsible Party: Sponsor
Other Study IDs: 14-071
Record Dates: First submitted 2014-04-10; First posted 2014-04-24 (Estimated); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer Survivors
Keywords: Treatment Exposure; Smoking History; 14-071

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, saliva or buccal sample for APOE analysis

GROUPS / COHORTS (3):
- breast cancer survivors who had received chemotherapy: Participants will complete all assessments at enrollment and approximately (+/- 16 weeks) at 8, 16, and 24 month follow-ups. We will screen participants to ensure that 50% of each group will report no smoking history and 50% will report a smoking history. Blood or buccal samples will be collected by trained staff one time at baseline. Those who choose not to provide the blood samples will be asked to provide a buccal sample as an alternative to test for APOE polymorphisms. Both patients and controls alive/deceased status will be tracked.
- breast cancer survivors who had not received chemotherapy: Participants will complete all assessments at enrollment and approximately (+/- 16 weeks) at 8, 16, and 24 month follow-ups. We will screen participants to ensure that 50% of each group will report no smoking history and 50% will report a smoking history. Blood or buccal samples will be collected by trained staff one time at baseline. Those who choose not to provide the blood samples will be asked to provide a buccal sample as an alternative to test for APOE polymorphisms. Both patients and controls alive/deceased status will be tracked.
- non-cancer controls matched by age,education, and race: Participants will complete all assessments at enrollment and approximately (+/- 16 weeks) at 8, 16, and 24 month follow-ups. We will screen participants to ensure that 50% of each group will report no smoking history and 50% will report a smoking history. Blood or buccal samples will be collected by trained staff one time at baseline. Those who choose not to provide the blood samples will be asked to provide a buccal sample as an alternative to test for APOE polymorphisms. Both patients and controls alive/deceased status will be tracked.

SUMMARY:
In this study,the investigators are looking to see how older women who are survivors of breast cancer and either did or did not receive chemotherapy are affected by treatment, compared to older women who have never had cancer. Thinking and memory abilities normally decrease with age and the investigators want to see if the long-term effects of cancer treatments may make these problems worse. The investigators will also look at how thinking and memory abilities of older women are affected by genetics and smoking history. Genetics and other factors may affect the brain's chemicals or structure, and may either protect against the negative effects on thinking or make someone more at risk for them.

MSK participants who previously consented to allostatic blood and saliva collection but have not yet provided any allostatic blood or saliva samples for this study, will not be asked to provide any further samples at follow-up. Participants who have consented to allostatic sample collection and provided one set of allostatic blood and saliva samples at a previous follow-up study visit will still be asked to provide a second set of samples at a later follow-up. COH participants will continue to provide allostatic blood and saliva collection as originally outlined

ELIGIBILITY:
Inclusion Criteria:

* The neuropsychological assessments were designed and validated in English and are not currently available in other languages. Translation of questionnaires into other languages would require reestablishing the reliability and validity of these measures. Therefore, participants must be able to communicate in English to complete the tests. Friend nominated, non-cancer controls will be frequency matched on age (+/- 5 years), education (less than college vs. some college and above), and race will be recruited using the same eligibility criteria as survivors except for no history of cancer.

For cancer patients, eligibility includes:

* As per medical record or self-report, post-menopausal female
* As per medical record or self-report, age 60 or older at recruitment
* As per medical record or self-report, age 55 or older at the time of breast cancer diagnosis
* As per medical record or self report, for cancers other than breast cancer or non-melanoma/basal cell skin cancer/squamous cell skin cancer:

  * Patient must be at least 3 years post diagnosis of that cancer
  * Not received chemotherapy treatment or external beam radiation for that cancer
* As per medical record or self-report, 5-15 years post diagnosis of breast cancer at the time of enrollment
* As per medical record or self-report, no evidence of any cancer disease
* American Joint Committee on Cancer (AJCC) stages 0-III breast cancer survivor as per clinical judgment/electronic medical record (EMR)
* Score of < 11 on the Blessed Orientation-Memory-Concentration Test (BOMC)
* In the judgment of the consenting professional, able to communicate well enough in English through verbal and written communication to complete the study assessments and provide informed consent

  * English proficiency verified through an adapted Bidimensional acculturation scale, score of 2.5 or above ***The scale will only be administered to participants who report also speaking a language other than English.

For controls participants, eligibility includes:

* As per medical record or self-report, post-menopausal female
* As per medical record or self-report, age 60 and older at recruitment
* In the judgment of the consenting professional, able to communicate well enough in English through verbal and written communication to complete the study assessments and provide informed consent

  °English proficiency verified through an adapted Bidimensional acculturation scale, score of 2.5 or above. ***The scale will only be administered to participants who report also speaking a language other than English.
* Score of < 11 on the Blessed Orientation-Memory-Concentration Test (BOMC)
* As per self report, no history of treatment with chemotherapy
* As per self report no history of cancer except non-melanoma/basal cell skin cancer squamous cell skin carcinoma

Exclusion Criteria:

* For cancer patients, exclusion criteria includes:

  * As per medical record or self report, diagnosis of neurodegenerative disorder that affects cognitive function (e.g., Alzheimer's, Parkinson's, Multiple Sclerosis, dementia, seizure disorders, etc)
  * As per medical record or self report, history of stroke or head injury requiring visit to the emergency room or hospitalization
  * As per medical record or self report, diagnosis of major Axis I psychiatric disorder including schizophrenia, manic-depressive disorder, or substance use disorders
  * As per self report or in the judgment of the consenting professional, visual or auditory impairment that would preclude ability to complete assessments
  * As per self report or as confirmed by the medical record, if the patient is taking anti-depression or anti-anxiety medication, < 2 months on these medication or a change in the prescribed dose in the past 2 months
  * Previously or actively participating in protocol MSK IRB# 10-079
* For control participants, exclusion criteria include

  * As per self report, diagnosis of neurodegenerative disorder that affects cognitive function (e.g., Alzheimer's, Parkinson's, Multiple Sclerosis, dementia, seizure disorders, etc.)
  * As per self report, history of stroke or head injury requiring visit to the emergency room or hospitalization
  * As per self report, diagnosis of major Axis I psychiatric disorder including schizophrenia, manic-depressive disorder, or substance use disorder
  * As per self report, or in the judgment of the consenting professional, visual or auditory impairment that would preclude ability to complete assessments
  * As per self report,if the person is taking anti-anxiety or anit-depression medication <2 months on these medications or a change in the prescribed dose in the past 2 months
  * Previously or actively participating in protocol 10-079

Min Age: 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We propose to enroll 540 participants into the study across the 2 sites: 270 participants (approximately 180 patients and 90 controls) from MSK and 270 participants from City of Hope (approximately 180 patients, and 90 controls).
Sampling Method: Non-Probability Sample
Enrollment: 499 (Actual)
Dates: Start 2014-04-08 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
neurocognitive outcomes | up to 24 months
  Neurocognitive tests will be performed longitudinally at 4 time points, enrollment, and 8, 16, and 24 months post enrollment.The participant will also be asked to complete two surveys.

CONTACTS AND LOCATIONS:
Overall Officials: James Root, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - City of Hope, Duarte, California
  - Memorial Sloan Kettering Cancer Center, New York, New York

REFERENCES:
- [Derived] Daniel E, Deng F, Patel SK, Sedrak MS, Kim H, Razavi M, Sun CL, Root JC, Ahles TA, Dale W, Chen BT. Brain white matter microstructural changes in chemotherapy-treated older long-term breast cancer survivors. Cancer Med. 2024 Jan;13(1):e6881. doi: 10.1002/cam4.6881. Epub 2023 Dec 28. PMID 38152038
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/